CLINICAL TRIAL: NCT07239219
Title: To Determine the Efficacy of Irrisept in Reducing Urinary Tract Infection During Urethral Catheter Removal.
Brief Title: The Impact of Irrisept in Reducing Urinary Tract Infection During Urethral Catheter Removal.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Principal Investigator, Hiren Patel, Assistant Professor, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20250670
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infection; Antibiotic; Catheter Infection
Keywords: UTI; antibiotic; Catheter infection; CAUTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — chlorhexidine gluconate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard of care
  Interventions: Other: Normal Saline
- Experimental (Experimental): Experimental
  Interventions: Other: 0.05% Chlorhexidine Gluconate

INTERVENTIONS:
Other: 0.05% Chlorhexidine Gluconate — 0.05% CHG is instilled into the bladder prior to trial of void.
  Arms: Experimental
Other: Normal Saline — Bladder is back filled with normal saline.
  Arms: Control

SUMMARY:
Given the high burden of post-catheter removal UTIs, this study aims to evaluate Irrisept instillation as a non-antibiotic intervention to reduce infection rates. By comparing Irrisept to saline irrigation, the study will provide critical insights into the efficacy of antiseptic bladder irrigation in preventing UTIs while minimizing antibiotic use. If successful, this approach could lead to new clinical guidelines for catheter removal protocols, improving patient outcomes and reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to the urology clinic for catheter removal
2. Must be 18 years or older.
3. The patient must be able to understand and willing to provide informed consent as described in this study protocol.
4. Must be willing to complete a post-catheter removal survey

Exclusion Criteria:

1. Allergy or adverse reaction to chlorohexidine gluconate
2. Under the age of 18
3. Refuse to provide informed consent
4. On antibiotic therapy for any indication.
5. Women who are pregnant or breastfeeding
6. Signs of skin or systemic infection
7. Patients undergoing catheter exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infection | 30 days
  Evaluate the rate of urinary tract infection after urethral catheter removal.

SECONDARY OUTCOMES:
Antibiotic use | 30 days
  Evaluate the rates of antibiotic use 30 days after urethral catheter removal
Adverse Events | 30 days
  Evaluate the rates of adverse events 30 days after urethral catheter removal

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided